CLINICAL TRIAL: NCT01165814
Title: Oral Naproxen Versus Oral Tramadol for Analgesia After Cesarean Delivery - A Randomized Controlled Trial
Brief Title: Naproxen Versus Tramadol for Post Cesarean Pain Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Ron Gonen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRAMNAP
Record Dates: First submitted 2010-07-18; First posted 2010-07-20 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Pain; Cesarean Section
Keywords: Pain control after cesarean section
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Tramadol at fixed intervals (Active Comparator)
  Interventions: Drug: Naproxen Tramadol
- Tramadol on request (Active Comparator)
  Interventions: Drug: Naproxen Tramadol
- Naproxen at fixed intervals (Active Comparator)
  Interventions: Drug: Naproxen Tramadol
- Naproxen on request (Active Comparator)
  Interventions: Drug: Naproxen Tramadol

INTERVENTIONS:
Drug: Naproxen Tramadol

SUMMARY:
Oral naproxen might be more efficacious for post-cesarean pain-control and have better side-effects profile than oral tramadol.

ELIGIBILITY:
Inclusion Criteria:

* all patients after cesarean section

Exclusion Criteria:

* emergent CS
* hypersensitivity to drug
* drug abuse

Sex: Female
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Pain Score

SECONDARY OUTCOMES:
Side effects

CONTACTS AND LOCATIONS:
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel